CLINICAL TRIAL: NCT06037291
Title: Assessment of the Soothing Effect of a Food Supplement on Sensitive and Reactive Skin. Double Blind Randomized Placebo-controlled Clinical Study.
Brief Title: Assessement of the Soothing Effect of a Food Supplement on Sensitive and Reactive Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT0002762/21
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coriander Seed Oil (Experimental): Dietary supplement - Coriander Seed Oil
  Interventions: Dietary Supplement: Coriander Seed Oil
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coriander Seed Oil — The study foresees the intake of 1 capsule per day during 56 days
  Arms: Coriander Seed Oil
Dietary Supplement: Placebo — The study foresees the intake of 1 capsule per day during 56 days
  Arms: Placebo

SUMMARY:
The study is aimed to assess the soothing effect of a food supplement composed of Coriander Seed Oil (CSO) in terms of reducing skin redness and skin discomfort (stinging feeling) on sensitive and reactive skin.

DETAILED DESCRIPTION:
A double blind, parallel groups, placebo-controlled study is carried out on 80 female subjects aged between 18 and 65 years old with sensitive and reactive skin.

The study foresees 56 days of products intake. Evaluations of the parameters under study are performed at baseline, after 14, 28 and 56 days of products consumption.

ELIGIBILITY:
Inclusion criteria :

* Good general health
* Caucasian ethnicity
* Female sex
* Phototype I to IV
* Sensitive and reactive skin (showing positive answer from 3-moderate to 4-strong to stinging test performed with a 10% lactic acid solution)
* Age between 18 and 65 years old (subject with 18 and 65 years old can be included)
* Subjects who have not been recently involved in any other similar study (evaluation is performed case by case by the experimenter but at least 1 month must be elapsed between a previous study on food supplement)
* Willingness to use during all the study period only the products to be tested
* Willingness not to use similar products that could interfere with the product to be tested
* Willingness to not vary the normal daily routine (i.e. lifestyle, physical activity, diet etc.)
* Subjects under effective contraception (oral/not oral) if women of childbearing potential; not expected to be changed during the trial
* Subject aware of the study procedures and having signed an informed consent form
* Subjects who accept not to expose in intensive way to UV rays during the whole study duration
* Subjects who have not involved in any sun test (for SPF evaluation) or tests that provide skin irradiation since less than two months

Exclusion Criteria:

* Subject does not meet the inclusion criteria,
* Pregnant/breastfeeding female or who have planned a pregnancy during the study period
* Subjects under systemically pharmacological treatment
* Subjects under locally pharmacological treatment on the skin area monitored during the test
* Subjects with congenital or acquired immunodeficiency
* Subjects under treatment with food supplements which could interfere with the functionality of the product under study
* Subjects which show skin alterations on the monitored area which could interfere with the functionality of the product under study
* Subjects considered as not adequate to participate to the study by the investigator
* Subjects with known or suspected sensitization to one or more test formulation ingredients
* Adult protected by law (under control or hospitalized in public or private institutions for reasons other than research, or incarcerated)
* Subjects not able to communicate or cooperate with the investigator for problems related to language, mental retardation or impaired brain function

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Skin redness | Baseline
  Induction of skin redness by skin stripping followed by the evaluation of skin color by CIELab color space (a* parameter)
Skin redness | 14 days
  Induction of skin redness by skin stripping followed by the evaluation of skin color by CIELab color space (a* parameter)
Skin redness | 28 days
  Induction of skin redness by skin stripping followed by the evaluation of skin color by CIELab color space (a* parameter)
Skin redness | 56 days
  Induction of skin redness by skin stripping followed by the evaluation of skin color by CIELab color space (a* parameter)

SECONDARY OUTCOMES:
Skin stinging | Baseline
  Induction of skin itching by a lactic acid solution followed by the self-assessment of stinging severity at different time points (0, 1, 2, 3, 4, 5, 7, 9, 12, 15 and 20 min) after the solution application using a defined 4-point clinical scale (1. No reaction; 2. Mild reaction; 3. Moderate reaction; 4. Severe reaction).
Skin stinging | 14 days
  Induction of skin itching by a lactic acid solution followed by the self-assessment of stinging severity at different time points (0, 1, 2, 3, 4, 5, 7, 9, 12, 15 and 20 min) after the solution application using a defined 4-point clinical scale (1. No reaction; 2. Mild reaction; 3. Moderate reaction; 4. Severe reaction).
Skin stinging | 28 days
  Induction of skin itching by a lactic acid solution followed by the self-assessment of stinging severity at different time points (0, 1, 2, 3, 4, 5, 7, 9, 12, 15 and 20 min) after the solution application using a defined 4-point clinical scale (1. No reaction; 2. Mild reaction; 3. Moderate reaction; 4. Severe reaction).
Skin stinging | 56 days
  Induction of skin itching by a lactic acid solution followed by the self-assessment of stinging severity at different time points (0, 1, 2, 3, 4, 5, 7, 9, 12, 15 and 20 min) after the solution application using a defined 4-point clinical scale (1. No reaction; 2. Mild reaction; 3. Moderate reaction; 4. Severe reaction).
Erythema index | Baseline
  Induction of skin redness by UVA+UVB exposure followed by the evaluation of the erythema index (skin haemoglobin content) by Mexameter® 24h after UV exposure.
Erythema index | 56 days
  Induction of skin redness by UVA+UVB exposure followed by the evaluation of the erythema index (skin haemoglobin content) by Mexameter® 24h after UV exposure.
Skin TNF-alpha quantification (subgroup of 20 subjects) | Baseline
  Quantification of TNF-alpha concentration by Enzyme-Linked Immunosorbent Assay on skin stripping performed 24h after UV exposure (non-irradiated and irradiated area)
Skin TNF-alpha quantification (subgroup of 20 subjects) | 56 days
  Quantification of TNF-alpha concentration by Enzyme-Linked Immunosorbent Assay on skin stripping performed 24h after UV exposure (non-irradiated and irradiated area)
Self-assessment of product efficacy | 56 days
  Questionnaire (10 questions with 4 possible answers : completely agree / agree / disagree / completely disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana De Ponti, Study Director — Complife Italia S.r.l
Locations (1):
- Complife Italia srl, Milan, Italy